CLINICAL TRIAL: NCT03235180
Title: Ultrasound Evaluation of Crohn's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to secure funding.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shiago Chen, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-001175
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Sulfur Hexafluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Crohn's Disease Subjects (Experimental): Subjects will receive ultrasound exams of the bowel with 2 different machines (Ultrasound Elastography and Ultrasound Vascularity) at three time points: baseline, 4 weeks, and 6 months. The ultrasound exams will be performed at first with no contrast agent, and then ultrasound measurements will be repeated with 1-2 ml of Sulfur Hexafluoride, a contract agent.
  Subjects also will receive Magnetic Resonance Enterography (MRE) exams at baseline and 6 months as part of their clinical care.
  Interventions: Drug: Sulfur Hexafluoride; Device: Ultrasound Elastography; Device: Ultrasound Vascularity; Device: Magnetic Resonance Enterography (MRE)

INTERVENTIONS:
Drug: Sulfur Hexafluoride — Subjects will receive ultrasound (US) imaging of the terminal ileum without and with sulfur hexafluoride contrast at baseline, 4 week and 6 months. Subjects will receive one to two milliliters of the contrast agent.
  Other Names: Lumason
Device: Ultrasound Elastography — Subjects will receive US Imaging with the GE Logiq E9 Ultrasound Scanner at baseline, 4 week and 6 months without and with contrast.
  Other Names: GE Logiq E9 Ultrasound Scanner
Device: Ultrasound Vascularity — Subjects will receive US Imaging with the Verasonics Ultrasound Scanner at baseline, 4 week and 6 months without and with contrast.
  Other Names: Verasonics
Device: Magnetic Resonance Enterography (MRE) — Subjects will receive MRE imaging at baseline and 6 months as part of regular clinical care.

SUMMARY:
The purpose of this study is to assess the effectiveness of a new ultrasound technology for evaluating Crohn's disease.

DETAILED DESCRIPTION:
The investigators will study the efficacy of ultrasound shear wave elastography and vascularity imaging for Crohn's Disease (CD) evaluation. Literature evidences demonstrate that bowel stiffness is correlated with fibrosis, while bowel vascularity and perfusion is correlated with inflammation. Therefore, the investigators expect the combination of shear wave elastography and vascularity imaging can increase the sensitivity and specificity of CD evaluation.

Ultrasound is safe, cost-effective, and widely accessible, thus provides an attractive alternative to the clinical standard Computed Tomography (CT), risks of radiation)) and Magnetic Resonance Imaging (MRI), more expensive and limited accessibility)).

Because ultrasound may not be able to image bowel loops deep in the body, its main role is for follow-up after initial screening by CT or MRI, especially for terminal ileum, which is easily accessible by ultrasound and the most frequently affected bowel segment for CD.

ELIGIBILITY:
Inclusion Criteria:

- Crohn's disease patients with involvement of terminal ileum (thickness > 3mm).

Exclusion Criteria:

* Patients with change of medicine or going to surgery over the 6-months follow-up period.
* Patients with unreliable ultrasound images due to conditions such as large body habitus or poor ultrasound imaging window.
* Adults lacking capacity to consent.
* Vulnerable subjects such as prisoners.
* Pregnant women and nursing mothers.
* Patients with known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunts.
* Patients with history of hypersensitivity allergic reactions to ultrasound contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigao Chen, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Crohn's Disease Subjects: Subjects will receive ultrasound exams of the bowel with 2 different machines (Ultrasound Elastography and Ultrasound Vascularity) at three time points: baseline, 4 weeks, and 6 months. The ultrasound exams will be performed at first with no contrast agent, and then ultrasound measurements will be repeated with 1-2 ml of Sulfur Hexafluoride, a contract agent.
  Subjects also will receive Magnetic Resonance Enterography (MRE) exams at baseline and 6 months as part of their clinical care.
  Sulfur Hexafluoride: Subjects will receive ultrasound (US) imaging of the terminal ileum without and with sulfur hexafluoride contrast at baseline, 4 week and 6 months. Subjects will receive one to two milliliters of the contrast agent.
  Ultrasound Elastography: Subjects will receive US Imaging with the GE Logiq E9 Ultrasound Scanner at baseline, 4 week and 6 months without and with contrast.
  Ultrasound Vascularity: Subjects will receive US Imaging with the Verasonics Ultrasound Scanner at baseline, 4 week and 6 months without and with contrast.
  Magnetic Resonance Enterography (MRE): Subjects will receive MRE imaging at baseline and 6 months as part of regular clinical care.
Period: Overall Study
Arm/Group | Crohn's Disease Subjects
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Crohn's Disease Subjects
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Shear Wave Speed
Description: Shear wave speed is a measure of small bowel stiffness; this will be measured on the General Electric (GE) Logiq E9 Ultrasound Scanner.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: KPa
Arm/Group | Crohn's Disease Subjects
Number analyzed (Participants) | 9
KPa | 8.42 (4.07)

2. Primary Outcome: Change in Vessel Density
Description: Vessel density is a measure of the vascularity of the bowel. It is the percentage of pixels in the bowel lesion with blood flow compared to the total area of the lesion. This will be measured with the Verasonics Ultrasound Scanner.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: percentage of pixels
Arm/Group | Crohn's Disease Subjects
Number analyzed (Participants) | 9
percentage of pixels | 14.1 (6.18)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 6 months on all participants.
Arm/Group | Crohn's Disease Subjects
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT03235180/Prot_SAP_000.pdf